CLINICAL TRIAL: NCT06310369
Title: Radiotherapy for BCG-unresponsive Non-muscle-invasive Carcinoma in Situ (CIS) Bladder Cancer: an Open-label, Single-arm, Multicenter, Phase 2 Study
Brief Title: Radiotherapy for BCG-unresponsive Non-muscle-invasive Carcinoma in Situ (CIS) Bladder Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EORTC 2335-GUCG
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Bladder Cancer
Keywords: NMIBC
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy arm (Experimental): Radiation therapy will be given covering the whole bladder over 4 weeks. The use of a radiosensitizing agent is mandatory.
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy — Radiation therapy will be given in 20 fractions of 2.75 Gy covering the whole bladder over 4 weeks.
  The use of a radiosensitizing agent is mandatory. Each recruiting center will have to choose 2 options of radiosensitizing agents.

SUMMARY:
The investigators aim to investigate a possible role for radiotherapy in good prognosis bladder cancer patients has been identified as a possible alternative to cystectomy, especially for patients non-eligible for surgery but has yet to be fully explored.

DETAILED DESCRIPTION:
Bladder cancer is the tenth most commonly diagnosed cancer with urothelial carcinoma representing 90% of all bladder cancer cases. Approximately three-quarters of patients diagnosed with urothelial carcinoma have non-muscle invasive disease (NMIBC) confined to the mucosa (stage Ta or carcinoma in situ (CIS)) or submucosa (stage T1). The gold standard for diagnosing CIS is a combination of cystoscopy, urine cytology, and histological evaluation. Diagnosis and resection of visible Ta/T1 tumors is done by transurethral resection of bladder tumors (TURBT). Standard treatment for patients with high-risk NMIBC (high-grade Ta, CIS, or any T1) following staging consists of intravesical Bacillus Calmette-Guerin (BCG) immunotherapy. BCG, even administered optimally, does not provide absolute protection. BCG failure is generally considered recurrence or progression during therapy. Clinical trial data comparing salvage therapies after BCG are quite heterogeneous, in part due to inconsistent definitions and reporting methods.

Patients who are BCG-unresponsive have a 20-40% risk for progression to muscle-invasive bladder cancer within 5 years, which carries a 50% risk for the development of incurable metastatic disease.

Interestingly, although chemoradiotherapy is a recognized standard of care in muscle-invasive bladder cancer (MIBC), it has not been adequately explored in NMIBC. However, the available data suggests that NMIBC is a radioresponsive malignancy and that in a proportion of patients bladder preservation would be possible.

The investigators aim to evaluate the use of radiotherapy in patients with high-grade non-muscle-invasive bladder cancer who have BCG failure, potentiating its effect with commonly use radiosensitizers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older with histologically confirmed, BCG-unresponsive, high-risk non-muscle-invasive bladder cancer of predominantly (>50%) urothelial histology who were ineligible for or declined to undergo radical cystectomy
* Patients with carcinoma in situ with or without high-grade Ta or T1
* Eastern Cooperative Oncology Group performance status of 0-2, and adequate organ function
* Patients with concomitant Ta and T1 tumours must have undergone complete TURBT, defined as per standard of care as a visually complete resection (residual carcinoma in situ, which is traditionally not amenable to complete transurethral resection is acceptable), and the most recent cystoscopy or TURBT must have been done within 12 weeks before study initiation. Presence of detrusor muscle on pathology samples is required to ensure sample adequacy. A second TURBT is recommended but not required for patients with T1 tumours. The use of either white-light cystoscopy or blue-light cystoscopy is permitted, but the same technique has to be used in a patient throughout the trial
* Definition of BCG unresponsive non-muscle-invasive bladder cancer according to the European Association of Urology (EAU) guidelines

Exclusion Criteria:

* Evidence of upper urinary tract carcinoma
* Hydronephrosis due to tumour in the presence of T1 disease
* Patients on current systemic therapy for bladder cancer
* Patients who have received pelvic external beam radiotherapy within the previous 5 years

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a complete response at 6 months post-radiotherapy | 6 months post-radiotherapy

SECONDARY OUTCOMES:
Progression-free survival | 5 years from randomisation
overall survival | 5 years from randomisation

CONTACTS AND LOCATIONS:
Overall Officials: Verane Achard, Dr, Study Chair — Fribourg Cantonal Hospital